CLINICAL TRIAL: NCT02306122
Title: Nudging Doctors to Collaborate With Pharmacists to Improve Medication Adherence
Brief Title: Pharmacy Home Adherence Reporting and Monitoring Outcomes Study
Acronym: PHARxMOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Tufts Medical Center (Other); Harvard University (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1010000295; 7RC4AG039072-02 (NIH)
Record Dates: First submitted 2014-11-02; First posted 2014-12-03 (Estimated); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Diabetes; Hypertension; Hypercholesterolemia
Keywords: medication adherence; choice architecture; pharmacy home
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Hypercholesterolemia; Medication Adherence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Default patient default doctor (Experimental): Patient nonadherence information sent to physician; Pharmacist calls patient unless physician cancels call
  Interventions: Behavioral: Pharmacist calls patient unless physician cancels call; Behavioral: Patient nonadherence information sent to physician
- Information patient default doctor (Experimental): Patient nonadherence information sent to physician
  Interventions: Behavioral: Patient nonadherence information sent to physician
- Control patient default doctor (No Intervention): Control - no intervention
- Choice patient choice doctor (Experimental): Patient nonadherence information sent to physician; Pharmacist calls patient if physician requests call
  Interventions: Behavioral: Patient nonadherence information sent to physician; Behavioral: Pharmacist calls patient if physician requests call
- Information patient choice doctor (Experimental): Patient nonadherence information sent to physician
  Interventions: Behavioral: Patient nonadherence information sent to physician
- Control patient choice doctor (No Intervention): Control - no intervention
- Information patient information doctor (Experimental): Patient nonadherence information sent to physician
  Interventions: Behavioral: Patient nonadherence information sent to physician
- Control patient information doctor (No Intervention): Control - no intervention
- Information doctor (Experimental): Physician receives nonadherence information, but there is no opportunity for pharmacist action
  Interventions: Behavioral: Doctor receives information and may be allowed certain actions
- Choice doctor (Experimental): Physician receives nonadherence information, and can choose to request pharmacist action
  Interventions: Behavioral: Doctor receives information and may be allowed certain actions
- Default doctor (Experimental): Physician receives nonadherence information; pharmacist action will be triggered unless physician cancels action
  Interventions: Behavioral: Doctor receives information and may be allowed certain actions

INTERVENTIONS:
Behavioral: Pharmacist calls patient unless physician cancels call
  Arms: Default patient default doctor
Behavioral: Patient nonadherence information sent to physician
  Arms: Choice patient choice doctor; Default patient default doctor; Information patient choice doctor; Information patient default doctor; Information patient information doctor
Behavioral: Pharmacist calls patient if physician requests call
  Arms: Choice patient choice doctor
Behavioral: Doctor receives information and may be allowed certain actions
  Arms: Choice doctor; Default doctor; Information doctor

SUMMARY:
This study is a pilot test of an intervention that delivers timely diagnostic information about medication nonadherence to doctors, and then offers the services of clinical pharmacists to treat these nonadherence problems. Participating doctors will be notified when a patient is 10 days late refilling a medication for diabetes, hypertension, or hypercholesterolemia. In one randomization arm the pharmacist will contact the patient as the default option (with no action required by the doctor), and in the other the pharmacist will contact the patient only if the doctor actively chooses that the pharmacist take action. Patients of participating doctors will be randomized to 1) one of these two pharmacist options, 2) an information only control arm in which the doctor gets adherence information but does not have access to a pharmacist for that patient, and 3) a no information control arm. The investigators' central hypothesis is that the pharmacist will be consulted more often when intervention by the pharmacist is the default outcome and that the default pharmacist intervention will be the most beneficial for adherence outcomes.

DETAILED DESCRIPTION:
Poor adherence with prescription medications is ubiquitous, regardless of the disease, medication, patient population, or country studied. It is also expensive - annual costs of poor adherence in the United States were recently estimated at $290 billion. This problem has two components: diagnosis and treatment. Regarding diagnosis, doctors' assessments of patients' adherence are inaccurate, and doctors often do not discuss adherence problems with their patients. This makes it attractive to use pharmacy claims to identify nonadherence. While diagnostic data is necessary to solve the non-adherence problem, it is not sufficient. Once diagnosed, doctors must take action to treat nonadherence. Research shows that simply giving doctors claims data about nonadherence is ineffective, probably because it is not clear what action to take, and because the costs in time and energy of taking action are too great. What is currently lacking is a practical way to effectively integrate this diagnostic information and treatment expertise into work flows in primary care doctors' offices, and an effective method of inducing doctors to act on it. Behavioral economics suggests that barriers to doctors' action may be overcome in a cost effective way by altering the architecture of choices doctors face.

The long term goal of this research is to develop systems that effectively connect pharmacy benefits managers (PBMs), primary care doctors, clinical pharmacists, and patients in ways that improve medication adherence and patients' health outcomes. The overall objective of this application, which is the next step toward attainment of the investigators long term goal, is to conduct a pilot test of an intervention that delivers timely diagnostic information about nonadherence to doctors, and then offers the services of clinical pharmacists to treat these nonadherence problems. Participating doctors will be notified when a patient is 10 days late refilling a medication for diabetes, hypertension, or hypercholesterolemia. Taking advantage of the principle of intelligent choice architecture from behavioral economics, in one arm the pharmacist will contact the patient as the default option (with no action required by the doctor), and in the other the pharmacist will contact the patient only if the doctor actively chooses that the pharmacist take action. Patients of participating doctors will be randomized to 1) one of these two pharmacist options, 2) an information only control arm in which the doctor gets adherence information but does not have access to a pharmacist for that patient, and 3) a no information control arm. The investigators central hypothesis, which is strongly supported by work in other fields, is that the pharmacist will be consulted more often when intervention by the pharmacist is the default outcome and that the default pharmacist intervention will be the most beneficial for adherence outcomes.

This study is a collaboration between researchers at Brown University, Tufts University, Harvard University, and Johns Hopkins University; Express Scripts; a large regional commercial insurer; and a network of primary care doctors in Eastern Massachusetts. The team is led by Dr. Ira Wilson, an experienced adherence researcher, and includes behavioral and health economists, and a statistician experienced in adherence issues. The investigators will accomplish the investigators overall objectives by pursuing the following Specific Aims:

1. Establish and test the technical and communications infrastructure required for the conduct of this clinical trial. The following steps must occur in a secure environment: a) Express Scripts notifies the study that a patient is late filling a prescription, b) the study notifies the doctor, c) the doctor makes a choice about how to respond, and d) a pharmacist, in some cases, contacts the patient.
2. Conduct and evaluate a clinical trial of an intervention comparing methods of offering pharmacist services to primary care doctors. Eligible doctors and patients will be randomized to a) pharmacist services under one of two choice architecture conditions (default or choice), b) adherence information only, or c) no information; further randomization for patients in the experimental arms will occur where the patient's HMO/PPO status will be revealed to the physician, or not. Outcomes include medication adherence, duration of nonadherence event, and physician participant behavioral outcomes.

ELIGIBILITY:
Physician Inclusion Criteria:

* New England Quality Care Alliance (NEQCA) primary care physicians of adult patients insured through large commercial insurer partner

Patient Inclusion Criteria:

* Adult patients of consented New England Quality Care Alliance (NEQCA) primary care physicians
* Insured through large commercial insurer partner
* Prescribed chronic medications for one or more of the three study conditions in the past six months

Patient Exclusion Criterion:

* On the insurer's "do not contact" list

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2697 (Actual)
Dates: Start 2011-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ira B Wilson, MD, MSc, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McConnell M, Rogers W, Simeonova E, Wilson IB. Architecting Process of Care: A randomized controlled study evaluating the impact of providing nonadherence information and pharmacist assistance to physicians. Health Serv Res. 2020 Feb;55(1):136-145. doi: 10.1111/1475-6773.13243. Epub 2019 Dec 13. PMID 31835278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Physician recruitment with signed consent forms was in-person. 91 physicians were consented and enrolled at launch. All eligible patients were automatically enrolled, and mailed an opt-out card to be returned if participation was refused.
Pre-assignment Details: Both patients and doctors were enrolled in the study. Separate Periods represent the sequential nature of the study design: Period 1 includes physicians only. Only those patients with a nonadherence event were randomized to a control or intervention arm, so the number consented at launch (2,606) is higher than the number included in the study results (1,474). Patients were removed if insurance coverage expired or if their enrolled physician withdrew.
Groups:
- Information Doctor: Physician randomized to Information Only arm
- Default Doctor: Physician randomized to Default arm
- Choice Doctor: Physician randomized to Choice arm
Period: Initial Physician Randomization
Arm/Group | Default Patient Default Doctor | Information Patient Default Doctor | Control Patient Default Doctor | Choice Patient Choice Doctor | Information Patient Choice Doctor | Control Patient Choice Doctor | Information Patient Information Doctor | Control Patient Information Doctor | Information Doctor | Default Doctor | Choice Doctor
Started (Patent participants are not included in this period.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29 | 31 | 31
Completed (Patient participants are not included in this period.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 28 | 31 | 31
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Post Nonadherence Subgroup Randomization
Arm/Group | Default Patient Default Doctor | Information Patient Default Doctor | Control Patient Default Doctor | Choice Patient Choice Doctor | Information Patient Choice Doctor | Control Patient Choice Doctor | Information Patient Information Doctor | Control Patient Information Doctor | Information Doctor | Default Doctor | Choice Doctor
Started (Only those patients with a nonadherence event are included in this period.) | 244 | 123 | 121 | 274 | 134 | 137 | 220 | 221 | 28 | 31 | 31
Completed | 244 | 123 | 121 | 274 | 134 | 137 | 220 | 221 | 28 | 31 | 31
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total is 1565, not 1564, because descriptive statistics were calculated for all physicians enrolled at randomization (91) rather than those enrolled at intervention (90)
Groups:
- Default Patient: Patient nonadherence information sent to physician; Pharmacist calls patient unless physician cancels call
- Information Patient: Patient nonadherence information sent to physician
- Control Patient: Control - no intervention
- Choice Patient: Patient nonadherence information sent to physician; Pharmacist calls patient if physician requests call
- Total: Total of all reporting groups
Arm/Group | Default Patient | Information Patient | Control Patient | Choice Patient | Information Doctor | Choice Doctor | Default Doctor | Total
Number analyzed (Participants) | 244 | 477 | 479 | 274 | 29 | 31 | 31 | 1565
Age, Continuous [Mean (Standard Deviation); unit: years] — years
  years | 56.80 (0.49) | 55.99 (0.51) | 56.58 (0.47) | 56.29 (0.68) | 53.86 (1.67) | 56.87 (1.53) | 56.16 (1.78) | 56.33 (0.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 167 | 163 | 107 | 16 | 11 | 12 | 554
  Male | 166 | 310 | 316 | 167 | 13 | 20 | 19 | 1011
Region of Enrollment [Number; unit: participants]
  United States | 244 | 477 | 479 | 274 | 29 | 31 | 31 | 1565

OUTCOME MEASURES:

1. Primary Outcome: Probability of Resolution of Nonadherence Within 30 Days
Description: Patients who were more than 10 days late refilling a chronic medication prescription were in the analytic sample frame and were targeted for intervention according to how they were randomized. This outcome is the rate at which these patients have filled a prescription by 30 days. Outcome is 1 if the patient fills the prescription by 30 days (considered resolution of nonadherence); otherwise it is 0. Outcome measures reported are the means of the per-person proportions of nonadherence (NAE) events resolved within 30 days across all patients in each particular arm.
Time Frame: Outcome measure examines fills within 30 days of a nonadherence event. Participants were followed over a total of 6 months.
Population: All Information Only patients are grouped together in these results (regardless of physician arm), because the treatment for all Information Only patients is identical across all physician arms.
Measure: Mean (Standard Deviation); unit: Proportion of resolved NAEs within 30
Groups:
- Control Patient: No information sent to physician, no opportunity for pharmacist intervention
Arm/Group | Default Patient | Choice Patient | Information Patient | Control Patient
Number analyzed (Participants) | 244 | 274 | 477 | 479
Proportion of resolved NAEs within 30 | .4286 (.4953) | .4290 (.4953) | .4554 (.4982) | .4437 (.4971)
Statistical Analysis 1: Comparison: Default Patient vs Control Patient; Test type: Superiority; p < 0.01, Regression, Logistic; Risk Difference (RD) = -0.015, Standard Error of Mean 0.034 — Comparator is control arm
Statistical Analysis 2: Comparison: Choice Patient vs Control Patient; Test type: Superiority; p < 0.01, Regression, Logistic; Risk Difference (RD) = -0.015, Standard Error of Mean 0.041 — Comparator is control arm
Statistical Analysis 3: Comparison: Information Patient vs Control Patient; Test type: Superiority; p < 0.01, Regression, Logistic; Risk Difference (RD) = 0.012, Standard Error of Mean 0.029 — Comparator is control arm

2. Primary Outcome: Duration of Nonadherence Event
Description: Patients who were more than 10 days late refilling a chronic medication prescription were in the analytic sample frame and were targeted for intervention according to how they were randomized. This outcome is the duration of nonadherence event (the length of time the patient took to refill a prescription if the refill had been late), in days.
Time Frame: Participants were followed over a total of 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Default Patient | Choice Patient | Information Patient | Control Patient
Number analyzed (Participants) | 244 | 274 | 477 | 479
Days | 40.91 (37.89) | 39.46 (35.02) | 41.35 (43.51) | 41.04 (41.80)
Statistical Analysis 1: Comparison: Default Patient vs Control Patient; Test type: Superiority; p < 0.01, Regression, Linear; Mean Difference (Final Values) = -0.128, Standard Error of Mean 2.523 — Comparator is the control arm
Statistical Analysis 2: Comparison: Choice Patient vs Control Patient; Test type: Superiority; p < 0.01, Regression, Linear; Mean Difference (Final Values) = -1.582, Standard Error of Mean 2.997 — Comparator is the control arm
Statistical Analysis 3: Comparison: Information Patient vs Control Patient; Test type: Superiority; p < 0.01, Regression, Linear; Mean Difference (Final Values) = 0.308, Standard Error of Mean 2.38 — Comparator is the control arm

3. Secondary Outcome: Probability of Physician Viewing Nonadherence Event Information
Description: Patients who were more than 10 days late refilling a chronic medication prescription were in the analytic sample frame and were targeted for intervention according to how they were randomized. This outcome is the rate at which physicians viewed nonadherence event information. Outcome measures reported are the means of the per-person proportions of NAE event notices viewed by the physician across all patients in each particular arm.
Time Frame: Participants were followed over a total of 6 months
Population: We excluded the Control group because we considered only claims where physicians assigned to a treatment arm would have been notified by email of nonadherence.
Measure: Mean (Standard Deviation); unit: Proportion of NAEs viewed
Groups:
- Information Only Patient: Patient nonadherence information sent to physician
Arm/Group | Default Patient | Choice Patient | Information Only Patient
Number analyzed (Participants) | 244 | 274 | 477
Proportion of NAEs viewed | 0.2822 (0.4505) | 0.3856 (0.4872) | 0.3257 (0.4688)
Statistical Analysis 1: Comparison: Default Patient vs Information Only Patient; Test type: Superiority; p < 0.01, Regression, Logistic; Risk Difference (RD) = -0.043, Standard Error of Mean 0.068 — Comparator is the information arm
Statistical Analysis 2: Comparison: Choice Patient vs Information Only Patient; Test type: Superiority; p < 0.01, Regression, Logistic; Risk Difference (RD) = 0.06, Standard Error of Mean 0.063 — Comparator is the information arm

4. Secondary Outcome: Probability of Pharmacist Action Triggered
Description: Patients who were more than 10 days late refilling a chronic medication prescription were in the analytic sample frame and were targeted for intervention according to how they were randomized. This outcome is the rate at which pharmacist action was triggered to resolve nonadherence. Outcome measures reported are the means of the per-person proportions of NAE events which triggered pharmacist action across all patients in each particular arm.
Time Frame: Participants were followed over a total of 6 months
Population: We considered only claims for patients who had been randomly assigned to intervention arms where the pharmacist was available - Default and Choice.
Measure: Mean (Standard Deviation); unit: Proportion with pharmacist calls
Arm/Group | Default Patient | Choice Patient
Number analyzed (Participants) | 244 | 274
Proportion with pharmacist calls | 0.6102 (0.4881) | 0.1903 (0.3929)
Statistical Analysis 1: Comparison: Default Patient vs Choice Patient; Test type: Superiority; p < 0.01, Regression, Logistic; Risk Difference (RD) = 0.42, Standard Error of Mean 0.071 — Comparator is the choice arm

ADVERSE EVENTS:
Time Frame: From launch of study to end of study (6 months)
Groups:
- Default Patient Default Doctor: Patient nonadherence information sent to physician; Pharmacist calls patient unless physician cancels call
  Pharmacist calls patient unless physician cancels call
  Patient nonadherence information sent to physician
- Choice Patient Choice Doctor: Patient nonadherence information sent to physician; Pharmacist calls patient if physician requests call
  Patient nonadherence information sent to physician
  Pharmacist calls patient if physician requests call
- Information Doctor; Choice Doctor; Default Doctor: Doctor receives information and may be allowed certain actions
Arm/Group | Default Patient Default Doctor | Information Patient Default Doctor | Control Patient Default Doctor | Choice Patient Choice Doctor | Information Patient Choice Doctor | Control Patient Choice Doctor | Information Patient Information Doctor | Control Patient Information Doctor | Information Doctor | Choice Doctor | Default Doctor
All-Cause Mortality (participants affected / at risk) | 0/244 | 0/123 | 0/121 | 0/274 | 0/134 | 0/137 | 0/220 | 0/221 | 0/29 | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/244 | 0/123 | 0/121 | 0/274 | 0/134 | 0/137 | 0/220 | 0/221 | 0/29 | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/244 | 0/123 | 0/121 | 0/274 | 0/134 | 0/137 | 0/220 | 0/221 | 0/29 | 0/31 | 0/31

LIMITATIONS AND CAVEATS:
We partnered with only one insurer and pharmacy benefit manager and therefore had information on adherence for a subset of any physician's patients. We only had information on selected medications. We could only track patient outcomes related to adherence. Few patients actually received the pharmacist intervention. A relatively high share of patients opted out of the research. Our multilevel experimental design, with randomization occurring at both patient and physician levels, was complex.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Informed Consent Form (2011-08-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT02306122/ICF_000.pdf